CLINICAL TRIAL: NCT01201915
Title: A Phase II, Multicenter, Open-label, Three-cohort Trial Evaluating the Efficacy and Safety of Vismodegib (GDC-0449) in Operable Basal Cell Carcinoma (BCC)
Brief Title: A Study Evaluating the Efficacy and Safety of Vismodegib (GDC-0449) in Operable Basal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHH4812g; GS01354 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2010-09-10; First posted 2010-09-15 (Estimated); Results first posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-05

CONDITIONS: Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — HhAntag691

ARMS (3):
- Cohort 1: Vismodegib 150 mg (Experimental): Participants received vismodegib 150 mg orally daily for 12 weeks.
  Interventions: Drug: Vismodegib
- Cohort 2: Vismodegib 150 mg (Experimental): Participants received vismodegib 150 mg orally daily for 12 weeks.
  Interventions: Drug: Vismodegib
- Cohort 3: Vismodegib 150 mg (Experimental): Participants received vismodegib 150 mg orally daily for 8 weeks, followed by 4 weeks with no treatment, followed by a second 8-week vismodegib treatment period.
  Interventions: Drug: Vismodegib

INTERVENTIONS:
Drug: Vismodegib — Vismodegib was supplied in gelatin capsules.
  Other Names: GDC-0449

SUMMARY:
This was a 3-cohort, open-label study of vismodegib (GDC-0449) in new (non-recurrent) operable basal cell carcinoma of the nodular subtype.

DETAILED DESCRIPTION:
For Cohort 1, the response to treatment was determined at the end of the 12 weeks of treatment. For Cohort 2, the response to treatment was determined after 12 weeks of treatment and 24 weeks of observation. For Cohort 3, the response to treatment was determined after intermittent dosing over a 20-week period, consisting of an initial 8-week treatment period, followed by a 4-week drug holiday period, followed by a second 8-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed new (not recurrent or previously treated) nodular basal cell carcinoma (BCC) at 1 of the listed anatomical sites, which must be biopsy confirmed at the study site.
* Willingness to consent to biopsy of the lesion.
* Willingness to delay excision of the target tumor site until the time mandated in the protocol, unless evidence of disease progression or lack of drug tolerability.
* Adequate hematopoietic capacity.
* Adequate hepatic function.
* For women of childbearing potential, agreement to use 2 acceptable forms of birth control (including one barrier method) during the study and for 7 months after discontinuation of study drug.
* For men with female partners of childbearing potential, agreement to use a male condom (with spermicide) and to advise their female partners to use an additional acceptable method of birth control during the study and for 2 months after discontinuation of study drug.
* Agreement not to donate blood/blood products during the study and for 7 months after discontinuing study drug.
* Agreement not to donate sperm or semen during treatment and for 2 months after the last dose of vismodegib.

Exclusion Criteria:

* Prior treatment with vismodegib or any Hedgehog pathway inhibitor.
* Inability or unwillingness to swallow capsules.
* Pregnancy or lactation.
* BCC with any clinical and histological pattern other than nodular BCC.
* Patients with known Gorlin's syndrome (basal cell nevus syndrome) or clinical suspicion of Gorlin's syndrome.
* Recent (ie, within the past 28 days), current, or planned participation in another experimental drug study.
* Use of any excluded medication or therapy within 21 days of study entry.
* History of other malignancies within 3 years of the first day of treatment (Day 1), except for tumors with a negligible risk of metastasis, such as other non-melanoma skin cancer (BCC, squamous cell cancer), ductal carcinoma in situ of the breast, or carcinoma in situ of the cervix.
* Uncontrolled medical illness.
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect interpretation of the results of the study or renders the patient at high risk for treatment complications.
* Any medical or psychological illness or condition preventing adequate consent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2010-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivor Caro, M.D., Study Director — Genentech, Inc.
Locations (12):
- United States (12):
  - Scottsdale, Arizona
  - Los Angeles, California
  - Redwood City, California
  - San Diego, California
  - St. Petersburg, Florida
  - Alpharetta, Georgia
  - Chicago, Illinois
  - Louisville, Kentucky
  - Philadelphia, Pennsylvania
  - Bartlett, Tennessee
  - Houston, Texas
  - Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1: Vismodegib 150 mg | Cohort 2: Vismodegib 150 mg | Cohort 3: Vismodegib 150 mg
Started | 24 | 25 | 25
Completed | 16 | 14 | 19
Not Completed | 8 | 11 | 6
Not completed — Adverse Event | 2 | 1 | 1
Not completed — Lost to Follow-up | 0 | 4 | 0
Not completed — Physician Decision | 3 | 0 | 0
Not completed — Subject Decision | 3 | 3 | 5
Not completed — Target Lesion Progression | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Treated participants population: All study participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Vismodegib 150 mg | Cohort 2: Vismodegib 150 mg | Cohort 3: Vismodegib 150 mg | Total
Number analyzed (Participants) | 24 | 25 | 25 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (11.2) | 65.2 (13.3) | 65.1 (11.8) | 63.6 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8 | 16
  Male | 19 | 22 | 17 | 58

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Histologic Clearance
Description: Complete histologic clearance was defined as the absence of histological evidence of basal cell carcinoma at the target tumor site. Histological examination was performed by an independent pathologist on specimens collected within 2 weeks of the end of treatment period, ie, at 12 weeks after Baseline in Cohort 1, at 36 weeks after Baseline in Cohort 2, and at 20 weeks after Baseline in Cohort 3.
Time Frame: Baseline to Week 12 (Cohort 1), Baseline to Week 36 (Cohort 2), Baseline to Week 20 (Cohort 3)
Population: Efficacy evaluable population: All participants who were treated with at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: Vismodegib 150 mg | Cohort 2: Vismodegib 150 mg | Cohort 3: Vismodegib 150 mg
Number analyzed (Participants) | 24 | 25 | 25
Percentage of participants | 42.0 [22.1 to 63.4] | 16.0 [4.5 to 36.1] | 44.0 [24.4 to 65.1]
Statistical Analysis 1: Comparison: Cohort 1: Vismodegib 150 mg; The null hypothesis was that percentage of participants with complete histologic clearance was 50% or less; Test type: Superiority or Other; p = 0.8463, 1-sided exact binomial test
Statistical Analysis 2: Comparison: Cohort 2: Vismodegib 150 mg; The null hypothesis was that percentage of participants with complete histologic clearance was 30% or less; Test type: Superiority or Other; p = 0.9668, 1-sided exact binomial test
Statistical Analysis 3: Comparison: Cohort 3: Vismodegib 150 mg; The null hypothesis was that percentage of participants with complete histologic clearance was 50% or less; Test type: Superiority or Other; p = 0.7878, 1-sided exact binomial test

2. Secondary Outcome: Time to Complete Clinical Clearance
Description: Time to complete clinical clearance was defined as the time from the first treatment with vismodegib until complete clinical clearance as determined by the investigator.
Time Frame: Baseline to the end of the study (up to 12 weeks for Cohort 1; up to 36 weeks for Cohort 2, up to 20 weeks for Cohort 3)
Population: Efficacy evaluable population: All participants who were treated with at least 1 dose of study drug. Only participants who achieved complete clinical clearance were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Cohort 1: Vismodegib 150 mg | Cohort 2: Vismodegib 150 mg | Cohort 3: Vismodegib 150 mg
Number analyzed (Participants) | 10 | 9 | 18
Days | 59.5 [28.0 to 80.0] | 84.0 [27.0 to 120.0] | 60.0 [55.0 to 86.0]

ADVERSE EVENTS:
Description: Safety population: All participants who were treated with at least 1 dose of study drug.
Arm/Group | Cohort 1: Vismodegib 150 mg | Cohort 2: Vismodegib 150 mg | Cohort 3: Vismodegib 150 mg
Serious Adverse Events (participants affected / at risk) | 0/24 | 3/25 | 3/25
Other Adverse Events (participants affected / at risk) | 24/24 | 25/25 | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Vismodegib 150 mg (N=24) | Cohort 2: Vismodegib 150 mg (N=25) | Cohort 3: Vismodegib 150 mg (N=25)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Vismodegib 150 mg (N=24) | Cohort 2: Vismodegib 150 mg (N=25) | Cohort 3: Vismodegib 150 mg (N=25)
Nausea (Gastrointestinal disorders) | 5 | 2 | 6
Constipation (Gastrointestinal disorders) | 0 | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 2
Fatigue (General disorders) | 5 | 3 | 7
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 3 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 3 | 0 | 4
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 19 | 19 | 18
Dysgeusia (Nervous system disorders) | 9 | 13 | 15
Ageusia (Nervous system disorders) | 10 | 5 | 7
Hypogeusia (Nervous system disorders) | 2 | 0 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 17 | 18
Madarosis (Skin and subcutaneous tissue disorders) | 3 | 2 | 3
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Hair Colour Changes (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3
Weight Decreased (Investigations) | 0 | 0 | 3
Influenza Like Illness (General disorders) | 0 | 0 | 2
Skin neoplasms malignant and unspecified (Excl melanoma) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.